CLINICAL TRIAL: NCT06632847
Title: Comparison of Inspiratory Muscle Training and Thera-band Resistive Training on Diaphragmatic Strength and Pulmonary Function of Healthy Adults.
Brief Title: Comparison of Device Based Inspiratory Muscle Training and Thera-band Resistive Training in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Umaila Rafique
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy Young Adults
Keywords: Inspiratory muscle training; Thera-band resistive training; Healthy young adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT with device (Experimental): IMT is a therapeutic approach designed to improve respiratory muscle strength and endurance. In this trail, participants will engage in a structured regimen of inspiratory exercises with high resistance.
  participants will perform inspiratory muscle exercises using the power-breathe device that provide intermediate to high resistance, with focus on both intensity and volume. The protocol involves 4 to 5 session per week.
  Interventions: Other: IMT based Resistance training
- Thera-band resistive training (Active Comparator): Participant will engage in a structured training that involving Thera-band resistance training. Participants use different color of thera-band that provides different resistance. The regimen includes 3 session per week using different colors of band.
  Interventions: Other: Theraband Resistive training

INTERVENTIONS:
Other: IMT based Resistance training — IMT with device group is trained twice daily, with the morning session and afternoon session. The intensity will increase progressively in this group, starting at 60% Maximal Inspiratory Pressure (MIP) and reaching 75% by the end of study. POSITION: Patient will be in sitting position. FREQUENCY: 4 TO 5 times per week. INTENSITY: 60 to 75% of MIP (gradually increment the load by 10%every 2 weeks to reach 75 to 80 %MIP). Time: 15 to 20 minutes.
  Arms: IMT with device
Other: Theraband Resistive training — IMT training is form of exercise designed to strengthen the muscle that are involve in inhalation, primarily the diaphragm and intercostal muscles. Thera-band resistive training perform twice daily, with morning and afternoon session. Training will be perform 3 times per week. POSITION: patient will be in standing position. INTENSITY: moderate intensity (black and green thera-band used to provide medium resistance). Time: 15 to 20 minutes
  Arms: Thera-band resistive training

SUMMARY:
This study aims to evaluate the impact of inspiratory muscle training and Thera-band resistive training on pulmonary function and diaphragmatic strength of healthy adults. This trail investigate whether IMT can improve pulmonary function and diaphragmatic strength of healthy adults as well as overall respiratory health.

DETAILED DESCRIPTION:
Inspiratory Muscle Training(IMT) has been shown to improve respiratory muscle strength and endurance in various conditions. This study aims to explore the effects of IMT specifically in healthy young adults. To assess whether a structured IMT program improves diaphragmatic strength and pulmonary function in healthy adults. A randomized control trail involving 56 competitive young healthy adults will be conducted. The study duration will be 8 weeks, with assessments conducted at baseline , mid-point, and at the end of intervention. The IMT group participate in 20 minutes of training session, 4 to 5 times per week, using power-breathe device. Thera-band resistive training group participate in 15 minutes of training session, 3 times per week, using different colors of thera-band. This study aims to provide robust evidence on the benefits of IMT for young healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants.
* 20 to 35 years
* FEV1/FVC ratio above 60%
* Non-smokers

Exclusion Criteria:

* Acute illness within last 2 weeks
* Obese patients whose BMI greater than 30kg
* Patient with history of chronic airflow limitation or any diagnosed disease.
* Patient with acute infection.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow Rate (PEFR) | 6 weeks
  peak expiratory flow rates measured through digital spirometer.3 zones of measurements are commonly used to interpret peak flow rates. Normal value of PEFR is 80 to 100%.Green zone indicates 80 to 100% normal peak flow reading, yellow zone indicates 50 to 79 %of normal peak flow readings, and red zone indicates less than 50% of normal peak flow reading.
Forced Vital Capacity (FVC) | 6 week
  Forced Vital Capacity (FVC) Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal. Changes in FVC from baseline to 3rd week and after 6 weeks day of intervention will be assessed.
Forced Expiratory volume in 1sec (FEV1) | 6 week
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, Phd, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Lazaro D, Corchete LA, Garcia JF, Jerves Donoso D, Lantaron-Caeiro E, Cobreros Mielgo R, Mielgo-Ayuso J, Gallego-Gallego D, Seco-Calvo J. Effects on Respiratory Pressures, Spirometry Biomarkers, and Sports Performance after Inspiratory Muscle Training in a Physically Active Population by Powerbreath(R): A Systematic Review and Meta-Analysis. Biology (Basel). 2022 Dec 29;12(1):56. doi: 10.3390/biology12010056. PMID 36671748
- [Background] Qin L, Liu S, Hu S, Feng L, Wang H, Gong X, Xuan W, Lu T. The Effect of Inspiratory Muscle Training on Health-Related Fitness in College Students. Int J Environ Res Public Health. 2024 Aug 17;21(8):1088. doi: 10.3390/ijerph21081088. PMID 39200697
- [Background] Van Hollebeke M, Gosselink R, Langer D. Training Specificity of Inspiratory Muscle Training Methods: A Randomized Trial. Front Physiol. 2020 Dec 3;11:576595. doi: 10.3389/fphys.2020.576595. eCollection 2020. PMID 33343384